CLINICAL TRIAL: NCT04410991
Title: A Phase 3, Randomized, Double-blind Efficacy and Safety Study Comparing SAR442168 to Teriflunomide (Aubagio®) in Participants With Relapsing Forms of Multiple Sclerosis
Brief Title: Relapsing Forms of Multiple Sclerosis (RMS) Study of Bruton's Tyrosine Kinase (BTK) Inhibitor Tolebrutinib (SAR442168) (GEMINI 2)
Acronym: GEMINI 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EFC16034; U1111-1238-1373 (Registry Identifier: ICTRP); 2020-000644-55 (EudraCT Number)
Record Dates: First submitted 2020-05-28; First posted 2020-06-01 (Actual); Results first posted 2025-06-18 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Relapsing Multiple Sclerosis
MeSH Terms: interventions — teriflunomide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SAR442168 (Experimental): Dose 1 of oral SAR442168 daily + placebo to match the teriflunomide tablet once daily
  Interventions: Drug: Tolebrutinib; Drug: Placebo to match Teriflunomide
- Teriflunomide (Active Comparator): Oral 14 mg oral teriflunomide + placebo to match the SAR442168 tablet once daily
  Interventions: Drug: Teriflunomide HMR1726; Drug: Placebo to match Tolebrutinib

INTERVENTIONS:
Drug: Tolebrutinib — Pharmaceutical form: Tablet
  Route of administration: Oral
  Other Names: SAR442168
  Arms: SAR442168
Drug: Teriflunomide HMR1726 — Pharmaceutical form: Tablet
  Route of administration: Oral
  Arms: Teriflunomide
Drug: Placebo to match Tolebrutinib — Pharmaceutical form: Tablet
  Route of administration: Oral
  Arms: Teriflunomide
Drug: Placebo to match Teriflunomide — Pharmaceutical form: Tablet
  Route of administration: Oral
  Arms: SAR442168

SUMMARY:
Primary Objective:

To assess efficacy of daily SAR442168 compared to a daily dose of 14 mg teriflunomide (Aubagio) measured by annualized adjudicated relapse rate (ARR) in participants with relapsing forms of MS

Secondary Objective:

To assess efficacy of SAR442168 compared to teriflunomide (Aubagio) on disability progression, MRI lesions, cognitive performance and quality of life To evaluate the safety and tolerability of daily SAR442168 To evaluate pharmacodynamics (PD) of SAR442168

DETAILED DESCRIPTION:
Study duration varied per participant in this event driven trial with a treatment duration of approximately 18 to 36 months. Participants completing the study were offered to participate in a long term safety study.

ELIGIBILITY:
Inclusion criteria :

* The participant must be 18 to 55 years of age, inclusive, at the time of signing the informed consent
* The participant must have been diagnosed with RMS according to the 2017 revision of the McDonald diagnostic criteria
* The participant has an expanded disability status scale (EDSS) score ≤5.5 at the first Screening Visit
* The participant must have at least 1 of the following prior to screening:

  * ≥1 documented relapse within the previous year OR
  * ≥2 documented relapses within the previous 2 years, OR
  * ≥1 documented Gd enhancing lesion on an MRI scan within the previous year
* Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies
* Male participants are eligible to participate if they agree to the following during the intervention period and until accelerated elimination procedure:

  * Refrain from donating sperm

Plus either:

* Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent OR
* Must agree to use contraception/barrier as detailed below
* Agree to use a male condom and should also be advised of the benefit for a female partner to use a highly effective method of contraception as a condom may break or leak when having sexual intercourse with a woman of childbearing potential (WOCBP) who is not currently pregnant

  - A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions apply:
* Is not a WOCBP OR
* Is a WOCBP and agrees to use a contraceptive method that is highly effective (with a failure rate of <1% per year), preferably with low user dependency during the intervention period and until accelerated elimination procedure is completed (or for at least 10 days after the last dose of SAR442168, if the case was unblinded) and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction during the study and for the same period of time.

  * A WOCBP must have a negative highly sensitive pregnancy test at screening and within 24hours before the first dose of study intervention.
  * If a urine test cannot be confirmed as negative (eg, an ambiguous result), a serum pregnancy test is required. In such cases, the participant must be excluded from participation if the serum pregnancy result is positive.
  * The Investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
  * The participant must have given written informed consent prior to undertaking any study related procedure. This includes consent to comply with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. In countries where the legal age of maturity is greater than 18 years, a specific ICF for such legally minor participants must also be signed by the participant's legally authorized representative

Exclusion criteria:

* The participant has been diagnosed with primary progressive multiplesclerosis (PPMS) according to the 2017 revision of the McDonald diagnostic criteria or with nonrelapsing secondary progressive multiplesclerosis (SPMS)
* The participant has a history of infection or may be at risk for infection including but not limited to: HIV, transplantation, live attenuated vaccines, progressive multifocal leukoencephalopathy, tuberculosis, hepatitis B or C, any persistent chronic or active recurring infection
* Clinically significant laboratory abnormalities (including evidence of liver injury) or electrocardiogram abnormalities at Screening.
* The participant has conditions or situations that would adversely affect participation in this study, including but not limited to:

  * A short life expectancy due to pre-existing health condition(s) as determined by their treating neurologist
  * Medical condition(s) or concomitant disease(s) making them nonevaluable for the primary efficacy endpoint or that would adversely affect participation in this study, as judged by the Investigator
  * A requirement for concomitant treatment that could bias the primary evaluation
* The participant has a history of or currently has concomitant medical or clinical conditions that would adversely affect participation in this study
* At screening, the participant is positive for hepatitis B surface antigen and/or hepatitis B core antibody and/or is positive for hepatitis C antibody
* The participant has any of the following:

  * A bleeding disorder or known platelet dysfunction at any time prior to the screening visit
  * A platelet count <150 000/μL at the screening visit
* The participant has a lymphocyte count below the lower limit of normal (LLN) at the screening visit
* The presence of psychiatric disturbance or substance abuse
* Prior/concomitant therapy
* The participant is receiving potent and moderate inducers of cytochrome P450 (CYP) 3A or potent inhibitors of CYP2C8 hepatic enzymes
* The participant is receiving anticoagulant/antiplatelet therapies
* The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 899 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2024-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (186):
- United States (43):
  - North Central Neurology Associates, PC-Site Number:8400009, Cullman, Alabama
  - Center for Neurology and Spine-Site Number:8400089, Phoenix, Arizona
  - Arcadia Neurology Center-Site Number:8400070, Arcadia, California
  - Multiple Sclerosis Center of California-Site Number:8400135, Newport Beach, California
  - Harbor UCLA-Site Number:8400088, Torrance, California
  - Mountain Neurological Research Center, Inc.-Site Number:8400128, Basalt, Colorado
  - Advanced Neurosciences Research-Site Number:8400025, Fort Collins, Colorado
  - South Florida Neurology Associates-Site Number:8400029, Boca Raton, Florida
  - University of Florida Health-Site Number:8400159, Gainesville, Florida
  - Neurology Associates, PA-Site Number:8400004, Maitland, Florida
  - University of Miami-Site Number:8400063, Miami, Florida
  - Infinity Clinical Research-Site Number:8400008, Sunrise, Florida
  - University of South Florida-Site Number:8400006, Tampa, Florida
  - Meridian Clinical Research-Site Number:8400003, Savannah, Georgia
  - Consultants In Neurology-Site Number:8400011, Northbrook, Illinois
  - Prairie Education and Research Cooperative-Site Number:8400071, Springfield, Illinois
  - Fort Wayne Neurological Center-Site Number:8400039, Fort Wayne, Indiana
  - CHI Saint Joseph Medical Group Neurology-Site Number:8400110, Lexington, Kentucky
  - University of Kentucky-Site Number:8400106, Lexington, Kentucky
  - Norton Neurology MS Services-Site Number:8400127, Louisville, Kentucky
  - The NeuroMedical Center-Site Number:8400057, Baton Rouge, Louisiana
  - International Neurorehabilitation Institute-Site Number:8400034, Lutherville-Timonium, Maryland
  - Wayne State University-Site Number:8400046, Detroit, Michigan
  - Minneapolis Clinic of Neurology-Site Number:8400051, Minneapolis, Minnesota
  - Saint Luke's Hospital-Site Number:8400153, Kansas City, Missouri
  - West Omaha Family Physicians-Site Number:8400139, Omaha, Nebraska
  - University Of Nebraska-Site Number:8400129, Omaha, Nebraska
  - Hackensack University Hospital-Site Number:8400047, Hackensack, New Jersey
  - University of New Mexico-Site Number:8400032, Albuquerque, New Mexico
  - South Shore Neurologic Associates-Site Number:8400100, Patchogue, New York
  - Novant Health Multiple Sclerosis Care Center - South Park-Site Number:8400120, Charlotte, North Carolina
  - Meridian Clinical Research, LLC-Site Number:8400005, Raleigh, North Carolina
  - Sanford Brain & Spine Center-Site Number:8400126, Fargo, North Dakota
  - Dayton Center for Neurological Disorders-Site Number:8400081, Centerville, Ohio
  - Jefferson Neurology Associates-Site Number:8400016, Philadelphia, Pennsylvania
  - Premier Neurology-Site Number:8400069, Greer, South Carolina
  - Advanced Neuroscience Center-Site Number:8400035, Franklin, Tennessee
  - Sibyl Wray, MD, Neurology, PC-Site Number:8400007, Knoxville, Tennessee
  - Mt Olympus Medical Research-Site Number:8400163, Katy, Texas
  - Neurology Center of San Antonio-Site Number:8400036, San Antonio, Texas
  - Texas Institute for Neuroogical Disorders-Sherman-Site Number:8400151, Sherman, Texas
  - Neurological Associates-Site Number:8400097, Richmond, Virginia
  - Wheaton Franciscan Healthcare-Site Number:8400022, Milwaukee, Wisconsin
- Argentina (5):
  - Investigational Site Number :0320004, CABA, Buenos Aires
  - Investigational Site Number :0320002, Capital Federal, Buenos Aires
  - Investigational Site Number :0320001, CABA, Buenos Aires F.D.
  - Investigational Site Number :0320003, Rosario, Santa Fe Province
  - Investigational Site Number :0320005, San Miguel de Tucumán
- Belgium (4):
  - Investigational Site Number :0560005, Bruges
  - Investigational Site Number :0560004, Ghent
  - Investigational Site Number :0560002, Mons
  - Investigational Site Number :0560001, Overpelt
- Brazil (3):
  - Investigational Site Number :0760001, Porto Alegre, Rio Grande do Sul
  - Investigational Site Number :0760002, Curitiba
  - Investigational Site Number :0760007, São Paulo
- Canada (6):
  - Investigational Site Number :1240002, Edmonton, Alberta
  - Investigational Site Number : 1240012, Hamilton, Ontario
  - Investigational Site Number :1240014, London, Ontario
  - Investigational Site Number :1240005, Greenfield Park, Quebec
  - Investigational Site Number :1240006, Gatineau
  - Investigational Site Number :1240021, Québec
- Chile (6):
  - Investigational Site Number :1520002, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number :1520005, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number :1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number :1520003, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number :1520006, Concepción
  - Investigational Site Number :1520004, Valdivia
- Croatia (3):
  - Investigational Site Number :1910001, Zagreb
  - Investigational Site Number :1910002, Zagreb
  - Investigational Site Number :1910003, Zagreb
- Czechia (5):
  - Investigational Site Number :2030002, Brno
  - Investigational Site Number :2030011, Hradec Králové
  - Investigational Site Number :2030001, Jihlava
  - Investigational Site Number :2030008, Prague
  - Investigational Site Number :2030005, Praha 5 - Motol
- France (12):
  - Investigational Site Number :2500019, Besançon
  - Investigational Site Number :2500018, Bordeaux
  - Investigational Site Number :2500011, Bron
  - Investigational Site Number :2500005, Clermont-Ferrand
  - Investigational Site Number :2500006, Montpellier
  - Investigational Site Number :2500010, Nantes
  - Investigational Site Number :2500002, Nice
  - Investigational Site Number :2500017, Nîmes
  - Investigational Site Number :2500007, Paris
  - Investigational Site Number :2500004, Poissy
  - Investigational Site Number :2500003, Rennes
  - Investigational Site Number :2500001, Strasbourg
- Germany (6):
  - Investigational Site Number :2760005, Bayreuth
  - Investigational Site Number :2760015, Berlin
  - Investigational Site Number :2760014, Berlin
  - Investigational Site Number :2760020, Bochum
  - Investigational Site Number :2760012, Essen
  - Investigational Site Number :2760003, Würzburg
- Greece (7):
  - Investigational Site Number :3000001, Athens
  - Investigational Site Number :3000006, Athens
  - Investigational Site Number :3000002, Athens
  - Investigational Site Number :3000007, Athens
  - Investigational Site Number :3000009, Athens
  - Investigational Site Number :3000004, Larissa
  - Investigational Site Number :3000003, Thessaloniki
- Hungary (4):
  - Investigational Site Number :3480105, Budapest
  - Investigational Site Number :3480102, Budapest
  - Investigational Site Number :3480106, Kaposvár
  - Investigational Site Number :3480103, Tatabánya
- India (5):
  - Investigational Site Number :3560005, Chandigarh
  - Investigational Site Number :3560007, Gūrgaon
  - Investigational Site Number :3560008, Gūrgaon
  - Investigational Site Number :3560002, New Delhi
  - Investigational Site Number :3560004, Thiruvananthapuram
- Israel (5):
  - Investigational Site Number :3760002, Ashkelon
  - Investigational Site Number :3760003, Haifa
  - Investigational Site Number :3760006, Rehovot
  - Investigational Site Number :3760004, Safed
  - Investigational Site Number :3760001, Tel Litwinsky
- Latvia (2):
  - Investigational Site Number :4280002, Riga
  - Investigational Site Number :4280003, Riga
- Investigational Site Number :5280001, Amsterdam, Netherlands
- Norway (2):
  - Investigational Site Number :5780002, Namsos
  - Investigational Site Number :5780001, Oslo
- Portugal (7):
  - Investigational Site Number :6200001, Braga
  - Investigational Site Number :6200005, Coimbra
  - Investigational Site Number :6200011, Lisbon
  - Investigational Site Number :6200006, Lisbon
  - Investigational Site Number :6200002, Matosinhos Municipality
  - Investigational Site Number :6200010, Porto
  - Investigational Site Number :6200004, Santa Maria da Feira
- San Juan MS Center-Site Number:8400015, Guaynabo, Puerto Rico
- Russia (12):
  - Investigational Site Number :6430006, Barnaul
  - Investigational Site Number :6430013, Bryansk
  - Investigational Site Number :6430001, Kazan'
  - Investigational Site Number :6430010, Kirov
  - Investigational Site Number :6430007, Moscow
  - Investigational Site Number :6430005, Moscow
  - Investigational Site Number :6430003, Novosibirsk
  - Investigational Site Number :6430014, Saint Petersburg
  - Investigational Site Number :6430004, Saint Petersburg
  - Investigational Site Number :6430002, Saint Petersburg
  - Investigational Site Number :6430011, Saransk
  - Investigational Site Number :6430012, Yekaterinburg
- Serbia (6):
  - Investigational Site Number :6880001, Belgrade
  - Investigational Site Number :6880003, Belgrade
  - Investigational Site Number :6880006, Belgrade
  - Investigational Site Number :6880002, Kragujevac
  - Investigational Site Number :6880004, Niš
  - Investigational Site Number :6880005, Novi Sad
- Slovakia (3):
  - Investigational Site Number :7030001, Bratislava
  - Investigational Site Number :7030002, Martin
  - Investigational Site Number :7030004, Nitra
- South Korea (4):
  - Investigational Site Number :4100001, Goyang-si, Gyeonggi-do
  - Investigational Site Number :4100003, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number :4100006, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number :4100002, Seoul, Seoul-teukbyeolsi
- Spain (13):
  - Investigational Site Number :7240011, Seville, Andalusia
  - Investigational Site Number :7240006, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number :7240009, Barakaldo, Bizkaia
  - Investigational Site Number :7240004, Salt, Girona [Gerona]
  - Investigational Site Number :7240013, Las Palmas de Gran Canaria, Las Palmas
  - Investigational Site Number :7240008, A Coruña
  - Investigational Site Number :7240007, L'Hospitalet de Llobregat
  - Investigational Site Number :7240005, Lleida
  - Investigational Site Number :7240003, Madrid
  - Investigational Site Number :7240001, Madrid
  - Investigational Site Number :7240002, Madrid
  - Investigational Site Number :7240010, Málaga
  - Investigational Site Number :7240012, Pozuelo de Alarcón
- Switzerland (3):
  - Investigational Site Number :7560003, Aarau
  - Investigational Site Number :7560002, Bern
  - Investigational Site Number :7560004, Lugano
- Turkey (Türkiye) (6):
  - Investigational Site Number :7920002, Ankara
  - Investigational Site Number :7920005, Besevler / Ankara
  - Investigational Site Number :7920006, Istanbul
  - Investigational Site Number :7920004, Kuttahta
  - Investigational Site Number :7920001, Samsun
  - Investigational Site Number :7920003, Trabzon
- Ukraine (9):
  - Investigational Site Number :8040020, Chernihiv
  - Investigational Site Number :8040002, Chernivtsi
  - Investigational Site Number :8040019, Chernivtsi
  - Investigational Site Number :8040005, Dnipro
  - Investigational Site Number :8040022, Kharkiv
  - Investigational Site Number :8040018, Kharkiv
  - Investigational Site Number :8040007, Kyiv
  - Investigational Site Number :8040006, Lviv
  - Investigational Site Number :8040003, Vinnytsia
- United Kingdom (3):
  - Investigational Site Number :8260003, Exeter, Devon
  - Investigational Site Number :8260016, Canterbury, Kent
  - Investigational Site Number :8260009, Bristol

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Oh J, Arnold DL, Cree BAC, Ionete C, Kim HJ, Sormani MP, Syed S, Chen Y, Maxwell CR, Benoit P, Turner TJ, Wallstroem E, Wiendl H; Tolebrutinib Phase 3 GEMINI 1 and 2 Trial Group. Tolebrutinib versus Teriflunomide in Relapsing Multiple Sclerosis. N Engl J Med. 2025 May 15;392(19):1893-1904. doi: 10.1056/NEJMoa2415985. Epub 2025 Apr 8. PMID 40202623
- See also: EFC16034 Plain language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25238&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 154 sites in 25 countries. A total of 1093 participants were screened from 11-Jun-2020 to 08-Aug-2022, of which 194 were screen failures. Screen failures were mainly due to not meeting eligibility criteria.
Pre-assignment Details: A total of 899 participants were randomized in this study in a 1:1 ratio to either teriflunomide 14 milligrams (mg) or tolebrutinib 60 mg group. This was an event-driven (6-month confirmed disability worsening [CDW]) trial with a variable treatment duration (end-of-study [EOS] duration: up to approximately 48 months).
Groups:
- Teriflunomide 14 mg: Participants received teriflunomide 14 mg tablet orally once daily (QD) along with a placebo matched to tolebrutinib orally QD up to approximately 48 months.
- Tolebrutinib 60 mg: Participants received tolebrutinib 60 mg tablet orally QD along with a placebo matched to teriflunomide orally QD up to approximately 46 months.
Period: Overall Study
Arm/Group | Teriflunomide 14 mg | Tolebrutinib 60 mg
Started | 452 | 447
Randomized and Treated | 451 | 447
Completed | 378 | 384
Not Completed | 74 | 63
Not completed — Poor compliance to protocol | 5 | 4
Not completed — Withdrawal by Subject | 59 | 55
Not completed — Other | 10 | 4

BASELINE CHARACTERISTICS:
Population: Analysis was performed on the randomized population.
Groups:
- Teriflunomide 14 mg: Participants received teriflunomide 14 mg tablet orally QD along with a placebo matched to tolebrutinib orally QD up to approximately 48 months.
- Total: Total of all reporting groups
Arm/Group | Teriflunomide 14 mg | Tolebrutinib 60 mg | Total
Number analyzed (Participants) | 452 | 447 | 899
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.1 (9.3) | 36.6 (9.3) | 36.4 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 293 | 300 | 593
  Male | 159 | 147 | 306
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 19 | 23 | 42
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 7 | 18
  White | 417 | 411 | 828
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Annualized Relapse Rate (ARR) as Assessed by Confirmed Protocol-defined Adjudicated Relapses
Description: Multiple sclerosis (MS) relapse was defined as a monophasic, acute or subacute onset of new neurological symptoms or worsening of previous neurological symptoms with an objective change on neurological examination. Symptoms were attributable to MS, lasted for >=24 hours with or without recovery, present at normal body temperature, and preceded by >=30 days of clinical stability.
Time Frame: Baseline (Day 1) to approximately 48 months
Population: The intent-to-treat (ITT) population included all randomized participants according to the intervention group allocated by the randomization, irrespective of the study intervention received.
Measure: Number (95% Confidence Interval); unit: relapses per participant year
Arm/Group | Teriflunomide 14 mg | Tolebrutinib 60 mg
Number analyzed (Participants) | 452 | 447
relapses per participant year | 0.109 [0.088 to 0.134] | 0.108 [0.089 to 0.131]
Statistical Analysis 1: Comparison: Teriflunomide 14 mg vs Tolebrutinib 60 mg; Analysis was performed using negative binomial model with number of adjudicated relapses onset between randomization date and EOS date as the response variable, treatment group, Gadolinium (Gd)-enhancing T1 lesions at baseline (presence, absence), expanded disability status scale (EDSS) strata (<4, >=4) and geographic region (United States [US], non-US) as covariates, and log transformed observation duration as the offset variable; Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error; p = 0.9758, Chi-squared — Threshold for significance at 2-sided 0.05 level; Relative risk = 0.996, 95% CI 2-sided [0.754 to 1.315]

2. Secondary Outcome: Time to Onset of 6-Month Confirmed Disability Worsening as Assessed by Expanded Disability Status Scale
Description: The EDSS was a disability scale that assessed the following 7 functional domains: visual, brainstem, pyramidal [motor], cerebellar [coordination], sensory, cerebral, and bowel/bladder. The total EDSS score ranged from 0 (normal) to 10 (death due to MS), increasing in increments of 0.5 points. Higher scores indicated increased disability. Time to onset of 6-month CDW was defined as the time from randomization to the onset of a confirmed, sustained increase from baseline in EDSS score (of >=1.5 points when the baseline score was 0, of >=1.0 point when the baseline score was 0.5 to <=5.5, of >=0.5 points when the baseline EDSS score was >5.5) over at least 6 months that was not attributable to another etiology.
Time Frame: Baseline (Day 1) to approximately 48 months
Population: The ITT population included all randomized participants according to the intervention group allocated by the randomization, irrespective of the study intervention received.
Measure: Median (Full Range); unit: months
Arm/Group | Teriflunomide 14 mg | Tolebrutinib 60 mg
Number analyzed (Participants) | 452 | 447
months | 12.14 [1.4 to 38.9] | 15.12 [2.0 to 37.1]
Statistical Analysis 1: Comparison: Teriflunomide 14 mg vs Tolebrutinib 60 mg; Analysis was performed using Cox proportional-hazards model with robust variance estimation. Covariates were treatment group, Gd-enhancing T1 lesions at baseline (presence, absence), EDSS strata (<4, >=4), geographic region (US, non-US); Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error; p = 0.0114, Log Rank — Derived from log-rank test with stratification of EDSS strata (<4, >=4), geographic region (US, non-US); Hazard Ratio (HR) = 0.582, 95% CI 2-sided [0.380 to 0.891]

3. Secondary Outcome: Time to Onset of 3-Month Confirmed Disability Worsening as Assessed by Expanded Disability Status Scale
Description: The EDSS was a disability scale that assessed the following 7 functional domains: visual, brainstem, pyramidal [motor], cerebellar [coordination], sensory, cerebral, and bowel/bladder. The total EDSS score ranged from 0 (normal) to 10 (death due to MS), increasing in increments of 0.5 points. Higher scores indicated increased disability. Time to onset of 3-month CDW was defined as the time from randomization to the onset of a confirmed, sustained increase from baseline in EDSS score (of >=1.5 points when the baseline score was 0, of >=1.0 point when the baseline score was 0.5 to <=5.5, of >=0.5 points when the baseline EDSS score was >5.5) over at least 3 months that was not attributable to another etiology.
Time Frame: Baseline (Day 1) to approximately 48 months
Population: as for outcome 2
Measure: Median (Full Range); unit: months
Arm/Group | Teriflunomide 14 mg | Tolebrutinib 60 mg
Number analyzed (Participants) | 452 | 447
months | 12.11 [1.4 to 39.1] | 12.11 [2.0 to 42.1]
Statistical Analysis 1: Comparison: Teriflunomide 14 mg vs Tolebrutinib 60 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error; p = 0.0181, Log Rank — Derived from log-rank test with stratification of EDSS strata (<4, >=4), geographic region (US, non-US); Hazard Ratio (HR) = 0.641, 95% CI 2-sided [0.444 to 0.925]

4. Secondary Outcome: Mean Number of New and/or Enlarging T2-Hyperintense Lesions Per Year
Description: Magnetic resonance imaging (MRI) of the brain was performed to identify number of new and/or enlarging T2-hyperintense lesions defined as the sum of the individual number of new and/or enlarging T2 lesions starting from baseline up to and including the EOS visit.
Time Frame: Baseline (Day 1) to approximately 48 months
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: number of new and/or enlarging T2lesions
Arm/Group | Teriflunomide 14 mg | Tolebrutinib 60 mg
Number analyzed (Participants) | 452 | 447
number of new and/or enlarging T2lesions | 4.369 [3.587 to 5.322] | 5.092 [4.340 to 5.975]
Statistical Analysis 1: Comparison: Teriflunomide 14 mg vs Tolebrutinib 60 mg; Analysis was performed using negative binomial model with the number of new and/or enlarging T2-hyperintense lesions between randomization date and EOS date as the response variable, treatment group, baseline T2-hyperintense lesion count, EDSS strata (<4, >=4) and geographic region (US, non-US) as covariates, and log transformed observation duration as the offset variable; Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error; p = 0.2362, Chi-squared; Relative risk = 1.165, 95% CI 2-sided [0.905 to 1.502]

5. Secondary Outcome: Mean Number of New Gadolinium-Enhancing T1-Hyperintense Lesions Per Scan
Description: MRI of the brain was performed to identify number of new Gd-enhancing T1-hyperintense lesions defined as the sum of the individual number of new Gd- enhancing T1-hyperintense lesions starting from baseline up to and including the EOS visit.
Time Frame: Baseline (Day 1) to approximately 48 months
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: number of new Gd-enhancing T1 lesions
Arm/Group | Teriflunomide 14 mg | Tolebrutinib 60 mg
Number analyzed (Participants) | 452 | 447
number of new Gd-enhancing T1 lesions | 0.217 [0.169 to 0.280] | 0.460 [0.365 to 0.581]
Statistical Analysis 1: Comparison: Teriflunomide 14 mg vs Tolebrutinib 60 mg; Analysis was performed using negative binomial model with the number of new Gd-enhancing T1-hyperintense lesions between randomization date and EOS date as the response variable, treatment group, Gd-enhancing T1 lesions at baseline (presence, absence), EDSS strata (<4, >=4) and geographic region (US, non-US) as covariates, and log transformed number of MRI scans as the offset variable; Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error; p < 0.0001, Chi-squared; Relative risk = 2.118, 95% CI 2-sided [1.502 to 2.987]

6. Secondary Outcome: Change From Baseline in Cognitive Function as Assessed by the Symbol Digit Modalities Test (SDMT) at EOS
Description: The SDMT was used to assess processing speed, divided attention, visual scanning, tracking and motor speed. It involved a simple substitution task using a reference key. The number of correct substitutions and number of items completed within a 90 second interval (maximum 110 seconds) were recorded. A decrease of 4 points from baseline on the SDMT was considered meaningful worsening. The score was the number of correctly coded items from 0-110 in 90 seconds; higher scores indicating a better outcome. Baseline was defined as the last available value prior to the first dose of study intervention.
Time Frame: Baseline (Day 1) to EOS (up to approximately 48 months)
Population: The ITT population included all randomized participants according to the intervention group allocated by the randomization, irrespective of the study intervention received. Only participants with data collected at specified timepoints are reported.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Teriflunomide 14 mg | Tolebrutinib 60 mg
Number analyzed (Participants) | 359 | 366
score on a scale | 0.428 (0.0373) | 0.374 (0.0370)
Statistical Analysis 1: Comparison: Teriflunomide 14 mg vs Tolebrutinib 60 mg; Covariates in the mixed-effect model with repeated measures (MMRM) were treatment group, EDSS strata (<4, >=4), geographic region (US, non-US), visit, treatment by visit interaction, baseline value, and baseline value-by-visit interaction; Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error; p = 0.3100, MMRM; Least square (LS) mean difference = -0.053, 95% CI 2-sided [-0.156 to 0.050]

7. Secondary Outcome: Change From Baseline in Cognitive Function as Assessed by the California Verbal Learning Test Second Edition (CVLT-II) at EOS
Description: The CVLT-II was a verbal learning and memory test consisting of recall and recognition of a list of 16 words. For each assessment, 5 trials were completed. Total Correct Recall Trials 1-5 was scaled to a normalized T-score metric, which had a mean of 50 and standard deviation of 10, the maximum possible score was 80 and a minimum was 0. Higher values indicated improved cognitive function. Baseline was defined as the last available value prior to the first dose of study intervention.
Time Frame: Baseline (Day 1) to EOS (up to approximately 48 months)
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Teriflunomide 14 mg | Tolebrutinib 60 mg
Number analyzed (Participants) | 347 | 357
T-score | 16.431 (0.6825) | 15.819 (0.6740)
Statistical Analysis 1: Comparison: Teriflunomide 14 mg vs Tolebrutinib 60 mg; Covariates in the MMRM were treatment group, EDSS strata (<4, >=4), geographic region (US, non-US), visit, treatment by visit interaction, baseline value, and baseline value-by-visit interaction; Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error; p = 0.5235, MMRM; LS mean difference = -0.612, 95% CI 2-sided [-2.493 to 1.269]

8. Secondary Outcome: Time to Onset of 6-Month Confirmed Disability Improvement (CDI) as Assessed by Expanded Disability Status Scale
Description: The EDSS was a disability scale that assessed the following 7 functional domains: visual, brainstem, pyramidal [motor], cerebellar [coordination], sensory, cerebral, and bowel/bladder. The total EDSS score ranged from 0 (normal) to 10 (death due to MS), increasing in increments of 0.5 points. Higher scores indicated increased disability. CDI was defined as a decrease of >=1 point from baseline in the EDSS score lasting at least 6 months.
Time Frame: Baseline (Day 1) to approximately 48 months
Population: as for outcome 2
Measure: Median (Full Range); unit: months
Arm/Group | Teriflunomide 14 mg | Tolebrutinib 60 mg
Number analyzed (Participants) | 452 | 447
months | 12.05 [2.8 to 30.6] | 9.04 [2.6 to 33.5]
Statistical Analysis 1: Comparison: Teriflunomide 14 mg vs Tolebrutinib 60 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error; p = 0.0079, Log Rank — Derived from log-rank test with stratification of EDSS strata (<4, >=4), geographic region (US, non-US); Hazard Ratio (HR) = 1.652, 95% CI 2-sided [1.145 to 2.383]

9. Secondary Outcome: Percent Change in Brain Volume Loss at EOS Compared to Month 6
Description: MRI of the brain was performed at the specified timepoints to detect the changes in brain volume loss.
Time Frame: Month 6 to EOS (up to approximately 48 months)
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Teriflunomide 14 mg | Tolebrutinib 60 mg
Number analyzed (Participants) | 307 | 317
percent change | -0.740 (0.0394) | -0.696 (0.0387)
Statistical Analysis 1: Comparison: Teriflunomide 14 mg vs Tolebrutinib 60 mg; Covariates in the MMRM were treatment group, EDSS strata (<4, >=4), geographic region (US, non-US), visit, treatment by visit interaction, cube root transformed Month 6 brain volume, and cube root transformed Month 6 brain volume-by-visit interaction; Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error; p = 0.4266, MMRM; LS mean difference = 0.044, 95% CI 2-sided [-0.065 to 0.153]

10. Secondary Outcome: Change From Baseline in Multiple Sclerosis Quality of Life 54 (MSQoL-54) Questionnaire Score at EOS
Description: MSQoL-54 was standardized instrument comprising generic and MS-specific items. This 54-item instrument generated 12 subscales and 2 single-item measures (satisfaction with sexual function [1 item]; change in health [1 item]). 12 subscales were: a: physical health (10 items), b: health perceptions (5 items), c: energy (5 items), d: role limit physical (4 items), e: sexual function (4 items), f: pain (3 items), g: social function (3 items), h: health distress (4 items), i: overall quality of life (2 items), j: emotional well-being (5 items), k: role limitations emotional (3 items) and l: cognitive function (4 items). Physical and mental health composite score were calculated as weighted sum of 'a to h' and 'i to l' subscales respectively. Each composite score was transformed linearly to common 0 (worst) to 100 (best) score range; higher score indicated improved quality of life. Baseline was defined as last available value prior to first dose of study intervention.
Time Frame: Baseline (Day 1) to EOS (up to approximately 48 months)
Population: The ITT population included all randomized participants according to the intervention group allocated by the randomization, irrespective of the study intervention received. Only participants with data collected at specified timepoints for the specified categories are reported.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Teriflunomide 14 mg | Tolebrutinib 60 mg
Number analyzed (Participants) | 357 | 370
score on a scale
  Physical health composite score: number analyzed (Participants) | 353 | 367
  Physical health composite score | -1.040 (0.7404) | -1.199 (0.7304)
  Mental health composite score | -1.657 (0.8709) | -1.390 (0.8581)

11. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Treatment-emergent Serious Adverse Events (TESAEs), TEAEs Leading to Permanent Study Intervention Discontinuation and Adverse Events of Special Interest (AESIs)
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. SAE was any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent disability/incapacity, was a congenital anomaly/birth defect or was an important medical event. An AESI was an AE (serious or nonserious) of scientific and medical concern specific to the Sponsor's product or program for which ongoing monitoring and immediate notification by the Investigator to the Sponsor was required. TEAEs were defined as AEs that developed, worsened or became serious during the treatment period.
Time Frame: From first dose of study intervention (Day 1) up to the earliest of either 10 days post last dose, death or last contact; up to approximately 48 months
Population: The safety population included all randomized participants exposed to the study intervention, regardless of the amount of exposure, analyzed according to the intervention actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Teriflunomide 14 mg | Tolebrutinib 60 mg
Number analyzed (Participants) | 451 | 447
Participants
  TEAEs | 387 | 385
  TESAEs | 37 | 49
  TEAEs leading to permanent study intervention discontinuation | 17 | 19
  TEAESIs | 40 | 46

12. Secondary Outcome: Change From Baseline in Plasma Neurofilament Light Chain (NfL) and Serum Chitinase-3 Like Protein-1 (Chi3L1) Levels at EOS
Description: Blood samples were collected at specified timepoints to assess change from baseline in NfL and Chi3L1. Baseline was defined as the last available value prior to the first dose of study intervention.
Time Frame: Baseline (Day 1) to EOS (up to approximately 48 months)
Population: The safety population included all randomized participants exposed to the study intervention, regardless of the amount of exposure, analyzed according to the intervention actually received. Only participants with data collected at specified timepoints for the specified categories are reported.
Measure: Median (Inter-Quartile Range); unit: picogram/milliliter
Arm/Group | Teriflunomide 14 mg | Tolebrutinib 60 mg
Number analyzed (Participants) | 311 | 319
picogram/milliliter
  NfL: number analyzed (Participants) | 301 | 314
  NfL | -0.900 [-4.390 to 0.770] | -0.150 [-3.560 to 2.750]
  Chi3L1 | -281.100 [-6148.400 to 5647.000] | 1462.500 [-4578.600 to 7002.700]

13. Secondary Outcome: Change From Baseline in Serum Immunoglobulin (Ig) Levels at EOS
Description: Blood samples were collected at specified timepoints to assess change from baseline in IgG and IgM levels. Baseline was defined as the last available value prior to the first dose of study intervention.
Time Frame: Baseline (Day 1) to EOS (up to approximately 48 months)
Population: as for outcome 12
Measure: Median (Inter-Quartile Range); unit: gram per liter
Arm/Group | Teriflunomide 14 mg | Tolebrutinib 60 mg
Number analyzed (Participants) | 281 | 287
gram per liter
  IgG | -0.590 [-1.330 to 0.230] | 0.140 [-0.720 to 1.060]
  IgM | -0.160 [-0.320 to -0.020] | -0.320 [-0.530 to -0.150]

ADVERSE EVENTS:
Time Frame: From first dose of study intervention (Day 1) up to the earliest of either 10 days post last dose, death or last contact; up to approximately 48 months. Deaths were collected from baseline (Day 1) up to end of follow-up, approximately 48 months.
Description: Analysis was performed on the safety population. All-cause mortality was performed on the randomized population. This was an event-driven (6-month CDW) trial with a variable treatment duration (EOS duration: up to approximately 48 months)
Arm/Group | Teriflunomide 14 mg | Tolebrutinib 60 mg
All-Cause Mortality (participants affected / at risk) | 2/452 | 1/447
Serious Adverse Events (participants affected / at risk) | 37/451 | 49/447
Other Adverse Events (participants affected / at risk) | 313/451 | 279/447
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teriflunomide 14 mg (N=451) | Tolebrutinib 60 mg (N=447)
Acute Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 3 (3) | 1 (1)
Bone Abscess (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Covid-19 (Infections and infestations) | 1 (1) | 2 (2)
Covid-19 Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Dengue Fever (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia Pyelonephritis (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 0 (0)
Gastroenteritis Norovirus (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia Aspiration (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Intraductal Proliferative Breast Lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oligodendroglioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous Cell Carcinoma Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Uterine Leiomyoma Necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Alcohol Withdrawal Syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Mental Fatigue (Psychiatric disorders) | 0 (0) | 1 (1)
Somatic Symptom Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide Attempt (Psychiatric disorders) | 0 (0) | 4 (4)
Facial Paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Generalised Tonic-Clonic Seizure (Nervous system disorders) | 0 (0) | 1 (2)
Guillain-Barre Syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Multiple Sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Multiple Sclerosis Relapse (Nervous system disorders) | 0 (0) | 1 (1)
Relapsing Multiple Sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Relapsing-Remitting Multiple Sclerosis (Nervous system disorders) | 0 (0) | 2 (2)
Trigeminal Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Vision Blurred (Eye disorders) | 1 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo Positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral Ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Duodenal Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis Acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bile Duct Stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug-Induced Liver Injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis Acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Calculus Urethral (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus Urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral Disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Abnormal Uterine Bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Adenomyosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Heavy Menstrual Bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Systemic Inflammatory Response Syndrome (General disorders) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 1 (1)
Transaminases Increased (Investigations) | 0 (0) | 1 (1)
Ankle Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gun Shot Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intentional Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint Dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament Rupture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ligament Sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon Rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal Burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teriflunomide 14 mg (N=451) | Tolebrutinib 60 mg (N=447)
Covid-19 (Infections and infestations) | 115 (131) | 106 (126)
Influenza (Infections and infestations) | 25 (35) | 27 (33)
Nasopharyngitis (Infections and infestations) | 64 (97) | 60 (102)
Upper Respiratory Tract Infection (Infections and infestations) | 36 (49) | 31 (43)
Urinary Tract Infection (Infections and infestations) | 30 (43) | 25 (35)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 24 (26) | 19 (28)
Neutropenia (Blood and lymphatic system disorders) | 34 (72) | 10 (14)
Anxiety (Psychiatric disorders) | 28 (33) | 24 (25)
Headache (Nervous system disorders) | 54 (64) | 61 (82)
Paraesthesia (Nervous system disorders) | 25 (30) | 16 (16)
Hypertension (Vascular disorders) | 34 (35) | 13 (14)
Diarrhoea (Gastrointestinal disorders) | 49 (57) | 22 (25)
Alopecia (Skin and subcutaneous tissue disorders) | 73 (74) | 37 (39)
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 (21) | 23 (35)
Back Pain (Musculoskeletal and connective tissue disorders) | 25 (39) | 27 (33)
Fatigue (General disorders) | 21 (22) | 30 (30)
Alanine Aminotransferase Increased (Investigations) | 23 (28) | 20 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2023-12-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT04410991/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT04410991/SAP_001.pdf